CLINICAL TRIAL: NCT05135286
Title: Multicenter, Double-Masked, Randomized, Safety and Efficacy Study of BRIMOCHOL™ PF and Carbachol PF Topical Ophthalmic Solution With Emmetropic Phakic and Pseudophakic Presbyopia
Brief Title: Safety and Efficacy Study of BRIMOCHOL™ PF and Carbachol PF in Subjects With Emmetropic Phakic and Pseudophakic Presbyopia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Visus Therapeutics (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VT-003
Record Dates: First submitted 2021-11-04; First posted 2021-11-26 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Presbyopia
MeSH Terms: conditions — Presbyopia | interventions — Carbachol; Brimonidine Tartrate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- BRIMOCHOL™ PF (Experimental): A single drop in each eye at a visit.
  Interventions: Drug: BRIMOCHOL™ PF
- Carbachol PF (Active Comparator): A single drop in each eye at a visit.
  Interventions: Drug: Carbachol PF
- Vehicle (Placebo Comparator): A single drop in each eye at a visit.
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: BRIMOCHOL™ PF — A single drop in each eye at a visit.
  Other Names: carbachol/brimonidine tartrate
  Arms: BRIMOCHOL™ PF
Drug: Carbachol PF — A single drop in each eye at a visit.
  Other Names: carbachol monotherapy
  Arms: Carbachol PF
Drug: Vehicle — A single drop in each eye at a visit.
  Arms: Vehicle

SUMMARY:
Safety and Efficacy Study of BRIMOCHOL™ PF and Carbachol PF in Subjects With Emmetropic Phakic and Pseudophakic Presbyopia

DETAILED DESCRIPTION:
Multicenter, Double-Masked, Randomized, Safety and Efficacy Study of BRIMOCHOL™ PF and Carbachol PF Topical Ophthalmic Solution With Emmetropic Phakic and Pseudophakic Presbyopia

ELIGIBILITY:
Inclusion Criteria:

* Male or female in good general health
* Must have presbyopia

Exclusion Criteria:

* History of allergic reaction to the study drug or any of its components
* Any disease or medical condition that, in the opinion of the Investigator, would prevent the subject from participating in the study or might confound study results

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 629 (Actual)
Dates: Start 2022-03-15 (Actual); Primary Completion 2025-03-13 (Actual); Study Completion 2025-03-13 (Actual)

PRIMARY OUTCOMES:
Change from baseline in near VA | Baseline Day 1
  Percentage of subjects with 3-line improvement in near VA without the loss of at least 1 line in distance VA

CONTACTS AND LOCATIONS:
Locations (42):
- United States (42):
  - Visus Therapeutics Investigative Site, Chandler, Arizona
  - Visus Therapeutics Investigative Site, Phoenix, Arizona
  - Visus Therapeutics Investigative Site, Sun City, Arizona
  - Visus Therapeutics Investigative Site, Glendale, California
  - Visus Therapeutics Investigative Site, Inglewood, California
  - Visus Therapeutics Investigative Site, Irvine, California
  - Visus Therapeutics Investigative Site, Mission Hills, California
  - Visus Therapeutics Investigative Site, Newport Beach, California
  - Visus Therapeutics Investigative Site, Pasadena, California
  - Visus Therapeutics Investigative Site, Santa Barbara, California
  - Visus Therapeutics Investigative Site, Littleton, Colorado
  - Visus Therapeutics Investigative Site, Danbury, Connecticut
  - Visus Therapeutics Investigative Site, Crystal River, Florida
  - Visus Therapeutics Investigative Site, Delray Beach, Florida
  - Visus Therapeutics Investigative Site, Fort Lauderdale, Florida
  - Visus Therapeutics Investigative Site, Jacksonville, Florida
  - Visus Therapeutics Investigative Site, Largo, Florida
  - Visus Therapeutics Investigative Site, Mt. Dora, Florida
  - Visus Therapeutics Investigative Site, Lake Villa, Illinois
  - Visus Therapeutics Investigative Site, Indianapolis, Indiana
  - Visus Therapeutics Investigative Site, Louisville, Kentucky
  - Visus Therapeutics Investigative Site, Bloomington, Minnesota
  - Visus Therapeutics Investigative Site, Kansas City, Missouri
  - Visus Therapeutics Investigative Site, St Louis, Missouri
  - Visus Therapeutics Investigative Site, Henderson, Nevada
  - Visus Therapeutics Investigative Site, Poughkeepsie, New York
  - Visus Therapeutics Investigative Site, Garner, North Carolina
  - Visus Therapeutics Investigative Site, West Fargo, North Dakota
  - Visus Therapeutics Investigative Site, Powell, Ohio
  - Visus Therapeutics Investigative Site, Portland, Oregon
  - Visus Therapeutics Investigative Site, Cranberry Township, Pennsylvania
  - Visus Therapeutics Investigative Site, Wilkes-Barre, Pennsylvania
  - Visus Therapeutics Investigative Site, Sioux Falls, South Dakota
  - Visus Therapeutics Investigative Site, Maryville, Tennessee
  - Visus Therapeutics Investigative Site, Memphis, Tennessee
  - Visus Therapeutics Investigative Site, Smyrna, Tennessee
  - Visus Therapeutics Investigative Site, Hurst, Texas
  - Visus Therapeutics Investigative Site, Lakeway, Texas
  - Visus Therapeutics Investigative Site, San Antonio, Texas
  - Visus Therapeutics Investigative Site, Draper, Utah
  - Visus Therapeutics Investigative Site, Falls Church, Virginia
  - Visus Therapeutics Investigative Site, Lynchburg, Virginia

IPD SHARING:
Plan to Share IPD: No